CLINICAL TRIAL: NCT00187200
Title: RESPONSE HF - Response of Cardiac Resynchronization Therapy Optimization With Interventricular (VV) Timing in Heart Failure Patients
Brief Title: Response of Cardiac Resynchronization Therapy Optimization With Ventricle to Ventricle Timing in Heart Failure Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRD299
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Results first posted 2015-09-25 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simultaneous VV Pacing (Active Comparator): Programmed to simultaneous biventricular pacing
  Interventions: Device: Simultaneous VV Pacing
- Sequential VV Pacing (Active Comparator): Programmed to sequential biventricular pacing
  Interventions: Device: Sequential VV Pacing

INTERVENTIONS:
Device: Simultaneous VV Pacing — Right ventricular and left ventricular pacing delivered simultaneously.
  Arms: Simultaneous VV Pacing
Device: Sequential VV Pacing — Right ventricular and left ventricular pacing delivered sequentially.
  Arms: Sequential VV Pacing

SUMMARY:
The purpose of the study is to evaluate the benefit of interventricular (V-V) delay optimization in reducing the non-responder rate in patients with cardiac resynchronization defibrillator (CRT-D) devices. The primary endpoint of this study is CRT responder rate.

For patients enrolled with new CRT-D systems, patients are considered non-responders if BOTH of the following requirements are fulfilled:

* < 10% improvement in 6-minute hall walk, and
* no class improvement or worsening in New York Heart Association (NYHA) scale.

For those receiving CRT-D devices as replacements of older CRT-D systems, patients are considered non-responders if BOTH of the following requirements are fulfilled:

* > 1 heart failure (HF) related hospitalization, and
* no class improvement or worsening in NYHA scale.

DETAILED DESCRIPTION:
Study Methods

* This is a prospective, randomized (simultaneous biventricular (BiV) pacing vs. sequential BiV pacing) study.
* Any patient that receives an FDA approved St. Jude Medical (SJM) CRT-D with V-V timing is eligible for enrollment.
* At 3 months post enrollment (or at implant for CRT-D replacements), patients screened as non-responders are randomized to either simultaneous or sequential BiV pacing. Patients requiring a replacement CRT-D device that are identified as non-responders to CRT are enrolled at the screening/randomization visit.
* Patients are followed for a period of 6 months post randomization:

  * Enrollment (1 week pre CRT-D implant to < 2 weeks post CRT-D implant)
  * Screening/Randomization Visit (3 months post enrollment)
  * Follow-up Visit (6 months post randomization)
* Total # of centers - 80 centers
* Sample size - 800 patients screened for CRT non-responders

ELIGIBILITY:
Inclusion Criteria:

* Patient has a standard indication for a CRT-D.
* Patient has the ability to complete a 6-minute hall walk with the only limiting factor to be fatigue or shortness of breath.
* Patient is geographically stable and willing to comply with the required follow-up schedule.
* Prior to 1 month of randomization, patient's HF medications are maintained stable and remain stable throughout the study.
* Patients requiring a CRT-D replacement must comply with BOTH of the following:

  * > 1 HF related hospitalization
  * No class improvement or worsening in NYHA scale

Exclusion Criteria:

* Patient's life expectancy is less than 12 months.
* Patient has had cardiac surgery within 6 months of enrollment.
* Patient has an epicardial ventricular lead system.
* Patient is less than 18 years old.
* Patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 816 (Actual)
Dates: Start 2005-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raul Weiss, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 816 patients were enrolled in the trial. Of the patients screened at the 3-month follow up, 572 patients were classified as responders and 102 patients as non-responders.
Pre-assignment Details: 102 of the patients were non-responders, but only 93 were randomized of which 57 completed the study and had data available for analysis. of the 816 participants screened only 93 wre randomized to treatment. This statement is accurate and appropriate.
Groups:
- Simultaneous Pacing V-V Timing: Patients maintained on simultaneous V-V delay
- Sequential VV Pacing: V-V delay was optimized
Period: Overall Study
Arm/Group | Simultaneous Pacing V-V Timing | Sequential VV Pacing
Started | 49 | 44
Completed | 31 | 26
Not Completed | 18 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simultaneous Pacing V-V Timing | Sequential VV Pacing | Total
Number analyzed (Participants) | 31 | 26 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 15 | 28
  >=65 years | 18 | 11 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (8.0) | 62.4 (11.2) | 65.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  United States | 31 | 26 | 57

OUTCOME MEASURES:

1. Primary Outcome: CRT Responder Rate
Description: Patients underwent baseline NYHA class and 6-minute hall walk distance (6-MHWD) assessment. After device implantation AV delays were optimized and all patients were programmed to simultaneous biventricular (BiV) pacing. At the 3-month follow-up, the NYHA class and 6-MHWD were reassessed. Non-responders were randomized 1:1 to either sequential BiV pacing with VV optimization or simultaneous BiV pacing. The responder rate at 6 months post randomization was compared between the two groups. Which is why the numbers are broken further down in the Outcome Measure table.
Time Frame: 6 months
Population: Per protocol analysis.
Measure: Number; unit: participants
Groups:
- Simultaneous Pacing V-V Timing: Patients maintained on simultaneous V-V delay per protocol
- Sequential VV Pacing: V-V delay was optimized per protocol
Arm/Group | Simultaneous Pacing V-V Timing | Sequential VV Pacing
Number analyzed (Participants) | 33 | 26
participants
  Responders | 16 | 20
  Non-Responders | 17 | 6

2. Secondary Outcome: NYHA Class Progression
Description: New York Heart Association (NYHA) functional classification provides a way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina pain.
Time Frame: 6 months
Population: Per protocol analysis
Measure: Number; unit: participants
Arm/Group | Simultaneous Pacing V-V Timing | Sequential VV Pacing
Number analyzed (Participants) | 30 | 26
participants
  NYYHA Class Improved by 1 category | 11 | 17
  NYHA Class Improved by more than 1 category | 1 | 1
  NYHA Class Unchanged | 17 | 7
  NYHA Class Worsened | 1 | 1

3. Secondary Outcome: 6 Minute Hall Walk Distance Test (6-MHWD)
Description: Patients were considered non-responders if the 6-MHWD had not improved by greater than or equal to 10% compared to baseline. This statement is accurate and appropriate.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Simultaneous Pacing V-V Timing | Sequential VV Pacing
Number analyzed (Participants) | 30 | 26
participants
  Responder | 10 | 13
  Non-Responder | 20 | 13

4. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Ejection fraction is a measurement of the percentage of blood leaving your heart each time it contracts. The left ventricle is the heart's main pumping chamber, so ejection fraction is usually measured only in the left ventricle (LV).
Time Frame: Randomization and 9 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Simultaneous Pacing V-V Timing | Sequential VV Pacing
Number analyzed (Participants) | 30 | 26
percentage
  Randomization | 30.6 (10.5) | 30.7 (10.5)
  9 Month Follow-up Visit | 32.6 (11.8) | 32.1 (11.6)

ADVERSE EVENTS:
Arm/Group | Simultaneous Pacing V-V Timing | Sequential VV Pacing
Serious Adverse Events (participants affected / at risk) | 8/31 | 2/26
Other Adverse Events (participants affected / at risk) | 7/31 | 12/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simultaneous Pacing V-V Timing (N=31) | Sequential VV Pacing (N=26)
ONSET OF ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
RV Lead Dislodgment or Migration (Cardiac disorders) | 1 (1) | 0 (0)
RV Elevated Pacing Thresholds (Cardiac disorders) | 1 (1) | 0 (0)
RV Decreased R/P-Wave Amplitude/Loss of Sensing (Cardiac disorders) | 1 (1) | 0 (0)
LEFT BRAIN TIA (Nervous system disorders) | 0 (0) | 1 (1)
LV Loss of capture (Cardiac disorders) | 1 (1) | 0 (0)
BACTEREMIA (Infections and infestations) | 0 (0) | 1 (1)
Therapy/Aborted Therapy for Non-Ventricular Rhythm:AF/AFL (Cardiac disorders) | 1 (1) | 0 (0)
MULTIPLE ICD FIRING, NSTEMI (Cardiac disorders) | 1 (1) | 0 (0)
CHEST PAIN AND AICD FIRING (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simultaneous Pacing V-V Timing (N=31) | Sequential VV Pacing (N=26)
DIAPHRAGMATIC CAPTURE BY ATRIAL LEAD (Cardiac disorders) | 1 (1) | 0 (0)
CHF EXACERBATION (Cardiac disorders) | 0 (0) | 1 (1)
CHF EXACERBATION + NEAR SYNCOPE (Cardiac disorders) | 0 (0) | 1 (1)
SHORTNESS OF BREATH (Cardiac disorders) | 0 (0) | 1 (1)
NEAR SYNCOPE WITH GENERAL WEAKNESS (Cardiac disorders) | 1 (1) | 0 (0)
HOSPITALIZATION FOR WEAKNESS WITH ICD FIRING X 2 (Cardiac disorders) | 0 (0) | 1 (1)
PNEUMONIA AND WORSENING KIDNEY FUNCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
END STAGE RENAL DZ - (WORSENING OF KNOWN DISEASE) (Renal and urinary disorders) | 0 (0) | 1 (1)
MRSA INFECTED LEFT ARM DIALYSIS GRAFT (Infections and infestations) | 0 (0) | 1 (1)
HOSPITALIZATION FOR NEAR SYNCOPE (Cardiac disorders) | 0 (0) | 1 (1)
DIZZY SPELL (General disorders) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ACUTE VIRAL PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1)
ABDOMINAL AORTIC ANEURYSM (Cardiac disorders) | 1 (1) | 0 (0)
SYNCOPE (Cardiac disorders) | 1 (1) | 0 (0)
SINUS INFECTION (General disorders) | 1 (1) | 0 (0)
COPD (CHRONIC) (Cardiac disorders) | 1 (1) | 0 (0)
EXACERBATION CONGESTIVE HEART FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
WORSENING RENAL FUNCTION (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the lower than expected non-responder rate at 3 months, the study did not reach the target randomized sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications and presentation should be presented to sponsor 30 days (manuscripts) or 7 days (abstracts) prior to submission for publication. The sponsor reserves the right to deny submission of study results if based on data owned by sponsor.